CLINICAL TRIAL: NCT00292019
Title: Robotic Laparoscopic Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-04-030; 10280
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Robotic prostatectomy: Patients who are eligible for a radical prostatectomy will have their surgery conducted with the aid of surgical robotics.
  Interventions: Procedure: Laparoscopic

INTERVENTIONS:
Procedure: Laparoscopic — Patients with prostate cancer who are eligible for a radical prostatectomy will have their surgery conducted with the aid of surgical robots.

SUMMARY:
This is a pilot study to evaluate the role of RALRP in the management of localized prostate cancer.

DETAILED DESCRIPTION:
To establish a robotic-assisted laparoscopic radical prostatectomy programme at the University of Western Ontario/London Health Sciences Centre and to critically evaluate the role of this programme in the management of localized prostate cancer in surgical candidates Details of surgical procedure, operative outcome, patient outcome including quality of life will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent
2. Locally confined, stage T1a, T2a or T2b prostate cancer
3. Aged 40-65 and judged by the study doctor to be a suitable candidate for a radical prostatectomy.
4. Serum prostate specific antigen equal to or less than 10mg/ml
5. Histologically confirmed adenocarcinoma of the prostate
6. Gleason score equal to or less than 7
7. Life expectancy of greater than 10 years.
8. Prostate size on TRUS measurement less than 40 grams

Exclusion Criteria:

1. Patients who have undergone prior hormone therapy.
2. Patients with a previous transurethral resectioning of the prostate (TURP)
3. History of other cancers other than basal cell carcinoma.
4. Patients with any prior abdominal surgery.
5. Any condition, or history of illness or surgery than, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient (eg significant cardiovascular conditions)
6. Patients with a large median lobe of the prostate. -

Exclusion Criteria:

-

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients eligible for a radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-03-04 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chin, MD< FRCSC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada